CLINICAL TRIAL: NCT06315127
Title: The CanDo (Canadian Donor Milk) Trial: Pasteurized Human Donor Milk Supplementation in the Well-baby Unit
Brief Title: The CanDo (Canadian Donor Milk) Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Mitacs (Industry)
Responsible Party: Principal Investigator, Sharon Unger, Principal Investigator, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-0119-A
Record Dates: First submitted 2023-11-10; First posted 2024-03-18 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Small for Gestational Age at Delivery; Gestational Diabetes; type1diabetes; Type2diabetes; Late Preterm Infant
Keywords: Donor milk; Exclusive breastfeeding; Infant health outcomes; Mother's milk; feed supplementation; late preterm infant; term infant
MeSH Terms: conditions — Diabetes, Gestational; Breast Feeding | interventions — Food, Formulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human Donor Milk (Experimental): All infants in this group will receive pasteurized donor milk from Rogers Hixon Ontario Human Milk Bank if they need extra feeding.
  Interventions: Dietary Supplement: Human donor milk
- Formula supplement (Active Comparator): All infants in this group will receive formula which is the standard of care if they need extra feeding.
  Interventions: Dietary Supplement: Formula

INTERVENTIONS:
Dietary Supplement: Human donor milk — The intervention will involve providing donor milk as required as a supplement to parent milk and will last for the duration of the infant's initial hospitalization. The intervention will continue throughout the hospitalization at any time that supplementation is recommended by the clinical team, and is expected to last from 0 to 72 hours post-birth. All donor milk will be aliquoted into individualized syringes in the Rogers Hixon Ontario Human Milk Bank which is located in Sinai Health. The decision regarding the timing and duration of the supplementation will be determined by the medical team in the well-baby unit based on the specific needs and circumstances of each mother-infant dyad. As this study follows a pragmatic approach, the clinical team will assess the need for supplementation based on the mother-infant dyad's condition.
  Other Names: Donor milk
  Arms: Human Donor Milk
Dietary Supplement: Formula — The intervention will involve providing formula as required as a supplement to parent milk and as a standard of care, and will last for the duration of the infant's initial hospitalization. The intervention will continue throughout the hospitalization at any time that supplementation is recommended by the clinical team, and is expected to last from 0 to 72 hours post-birth. The formula will be supplied from the hospital's inventory in accordance with the standard procedure followed by the well-baby unit to supplement infants. The decision regarding the timing and duration of the supplementation will be determined by the medical team in the well-baby unit based on the specific needs and circumstances of each mother-infant dyad.
  Other Names: Cow's milk based formula
  Arms: Formula supplement

SUMMARY:
The goal of this clinical trial is to learn about the impact of donor milk vs formula supplementation on human milk feeding and the health outcomes of infants who require supplementation in well-baby units. It aims to explore whether supplementation with donor milk vs formula for infants during the initial hospital stay in a well-baby unit will increase both the exclusivity and duration of breastfeeding at 4 months. The Investigators will also explore whether the type of supplementation will positively affect measures of newborns' health, growth, behavior, feeding efficacy, and parental stress. Each participating infant born to a diabetic mother OR born small for his/her gestational age (<2500 grams) OR late preterm (35 0/7-36 6/7 weeks of gestational age) is assigned at random to 2 groups. The groups are: 1) Donor milk: all babies in this group will receive pasteurized donor milk from a trusted milk bank. 2) Formula: all babies in this group will receive formula as a standard of care.

DETAILED DESCRIPTION:
Background and Importance: Human milk is the ideal nutrition for all infants, and research has demonstrated that human donor milk can provide health benefits for preterm infants. Approximately 35-50% of late preterm and term infants admitted to a well-baby unit after birth require supplementation due to various reasons including hypoglycemia, weight loss, or insufficient availability of parent's milk. However, there is limited research to guide decision making on which supplement to prescribe. Despite this, many hospitals are introducing donor milk in well-baby units in light of the growing recognition of the health protective effects of human milk.

Goals/ Research Aims: The primary research aim of this study is to compare the effects of supplementing parent's milk with donor milk versus formula in infants at increased risk for supplementation (infant born to a mother with diabetes, infant with a birth weight smaller than expected for the gestational age (SGA)) on exclusive human milk feeding at 4 months of age. Secondary research aims include: examining the effects of supplementing parent's milk with donor milk on any or exclusive human milk feeding rates at 1, 2 and 3 months, infant health and growth at hospital discharge and at 1, 2, 3, and 4 months, and breast feeding self-efficacy scores. Exploratory outcomes include: infant temperament scores at 1, 2, 3, and 4 months, and parental mental health scores at 2 and 4 months using validated questionaires, milk cortisol concentrations at 2 and 4 months, the use of informally shared milk, and the associated financial costs of a donor milk program versus formula.

Methods/ Approaches/ Expertise: This proposed study is a randomized, controlled, single-center trial that will involve assigning participants to two intervention arms (n=56 infants/arm). The intervention will involve providing donor milk or formula in bottles and will last for the duration of the infant's initial hospitalization, followed by monthly phone calls and a virtual or in-person assessment at 4 months. At each time-point of 1, 2, 3, and 4-month, surveys of breast feeding self-efficacy, and health and infant temparement will be conducted, and the infant's anthropometrics will be measured. Additionally, measures of parental depression, anxiety and stress will be assessed with survey-based tools at 2 and 4 months. A coincident human milk sample will be collected at 2 and 4 months and will be analysed for cortisol concentrations. The research team has experience running feeding interventions and donor milk trials in newborns, and includes experts in nursing, medicine, dietetics, and milk banking.

Expected Outcomes: This proposed research holds the potential to make a meaningful impact on public health. In Canada, with approximately 350,000 level I nursery admissions each year and high rates of formula supplementation ranging from 35-50%, there is a clear opportunity for improvement. By promoting exclusive human milk feeding, exploring evidence-based practices to inform hospital guidelines, and reducing the reliance on informal milk sharing, this research aims to enhance the health outcomes for both parents and infants. Additionally, it seeks to deepen the understanding of early parent-child interactions, fostering greater awareness and knowledge in this area.

ELIGIBILITY:
Inclusion Criteria:

Infants admitted to the well-baby unit at Sinai Health whose parent(s) intend to feed parent milk and who require supplementation:

* Infants of gestational/ type 1/ type 2 diabetic mothers
* Infants who are born small for gestational age (SGA) by using a sex-specific reference population and determining if their birth weight falls below the 10th percentile for gestational age
* Infants with a birth weight less than 2.5 kg
* Late preterm infants born between 35 0/7-36 6/7 weeks of gestational age

Exclusion Criteria:

* Enrollment in any other clinical study affecting nutritional management during the feeding intervention; anticipated change in primary caregiver (person providing the feed) prior to 4 months; refusal to consent to donor milk; supplementation with formula prior to enrollment; any physical condition that may impact growth (ex: skeletal dysplasia).

Max Age: 2 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Donor milk supplementation and exclusive breastfeeding rate at 4 months | At 4 months follow up
  To determine whether the provision of donor milk as prescribed as a supplement to parent's milk for infants at higher risk for supplementation and admitted to a well-baby unit improves exclusive human milk feeding rate at 4 months of age compared to supplementation with formula.

SECONDARY OUTCOMES:
Exploring donor milk supplementation and exclusive or any breastfeeding rate at 1, 2, and 3 months | At 1, 2, and 3 months follow ups
  To determine whether the provision of donor milk as prescribed as a supplement to parent's milk for infants at higher risk for supplementation and admitted to a well-baby unit improves any, or exclusive, human milk feeding rates at 1, 2, and 3 months of age rate compared to supplementation with formula.
Exploring donor milk supplementation and breastfeeding self-efficacy scores at 1, 2, 3 and 4 months | At 1, 2, 3, and 4 months follow ups
  To determine whether the provision of donor milk as prescribed as a supplement to parent's milk for infants at higher risk for supplementation and admitted to a well-baby unit improves breastfeeding self-efficacy scores at 1, 2, 3, and 4 months compared to supplementation with formula. Breastfeeding Self-Efficacy Scale - Short Form, BSES-SF will be used which consists of 14 items scored on a 5-point Likert scale ranging from not at all confident to always confident. Individuals who score higher on the BSES-SF are expressing more confidence in their ability to breastfeed successfully.
Exploring donor milk supplementation and glucose concentrations during hospital stay | From 2 to 72 hours after delivery or until discharge
  To determine whether the provision of donor milk as prescribed as a supplement to parent's milk for infants at higher risk for supplementation and admitted to a well-baby unit improves hypoglycemia in infants compared to supplementation with formula. Glucose concentrations during hospital stay and at discharge will be extracted from patient charts and compared between groups.
Exploring donor milk supplementation and percent weight loss during hospital stay | From birth to 72 hours after delivery or until discharge.
  To determine whether the provision of donor milk as prescribed as a supplement to parent's milk for infants at higher risk for supplementation and admitted to a well-baby unit improves weight loss in infants compared to supplementation with formula. Infant weight during the hospital stay and at discharge will be extracted from patient charts and percent weight loss will be compared between groups.
Exploring donor milk supplementation and the length of hospital stay | From birth to 72 hours after delivery or until discharge
  To determine whether the provision of donor milk as prescribed as a supplement to parent's milk for infants at higher risk for supplementation and admitted to a well-baby unit affects their length of hospital stay compared to supplementation with formula.
Exploring donor milk supplementation and weight measurements | 1, 2, 3, and 4 months
  To determine whether the provision of donor milk as prescribed as a supplement to parent's milk for infants at higher risk for supplementation and admitted to a well-baby unit affects their weight compared to supplementation with formula at 1, 2, 3, and 4 months using standardized procedures including mechanical scales.
Exploring donor milk supplementation and length measurements | 1, 2, 3, and 4 months
  To determine whether the provision of donor milk as prescribed as a supplement to parent's milk for infants at higher risk for supplementation and admitted to a well-baby unit affects their length compared to supplementation with formula at 1, 2, 3, and 4 months using standardized procedures including length boards.
Exploring donor milk supplementation and head circumference measurements | 1, 2, 3, and 4 months
  To determine whether the provision of donor milk as prescribed as a supplement to parent's milk for infants at higher risk for supplementation and admitted to a well-baby unit affects their head circumference compared to supplementation with formula at 1, 2, 3, and 4 months using standardized procedures including non-stretchable measuring tapes.

OTHER OUTCOMES:
Exploratory outcome: exploring donor milk supplementation and infant temperament scores | 1, 2, 3 and 4 months
  To explore whether the provision of donor milk as a supplement to parent's milk affects infant temperament scores at 1, 2, 3, and 4 months compared to supplementation with formula using validated questionnaire called Infant Behavior Questionnaire-Revised, Very Short Form which is a survey of 37 items spanning 3 broad scales including negative emotionality, positive affectivity, and orienting/ regulatory capacity. In this questionnaire, a high score indicates a greater degree of the respective characteristic being measured. For example, a high score in negative emotionality suggests a higher frequency or intensity of negative emotions, while a high score in positive affectivity indicates a greater expression of positive emotions. Similarly, a high score in orienting/regulatory capacity suggests better attentional control and regulatory abilities in the infant.
Exploratory outcome: exploring donor milk supplementation and parent's anxiety | 2 and 4 months
  To explore whether the provision of donor milk as a supplement to the parent's milk affects the parent's mental health. Anxiety will be measured with the State-Trait Anxiety Inventory (STAI) which has been used to assess trait (20 items) and state (20 items) anxiety. STAI has been used to differentiate anxiety from depressive syndromes and to generally assess caregiver distress in research. A high score on either the trait or state anxiety scale of the STAI suggests a greater degree of anxiety experienced by the individual being assessed.
Exploratory outcome: exploring donor milk supplementation and parent's depression | 2 and 4 months
  To explore whether the provision of donor milk as a supplement to parent's milk affects parent's mental health at 2 and 4 months using a validated questionnaire called The Edinburgh Postnatal Depression Scale (EPDS). This questionnaire has been classically described for screening for postpartum depression in mothers using a 10-point scale. Typically, cutoff scores are used to classify individuals as at risk for postpartum depression, with higher scores indicating a higher risk level.
Exploratory outcome: exploring donor milk supplementation and maternal cortisol concentrations | 2 and 4 months
  To explore whether the provision of donor milk as a supplement to parent's milk affects maternal cortisol concentrations at 2, and 4 months. Timed milk samples (morning sample to account for diurnal variation) will be collected at 2 and 4 months of age. These samples will be collected in the morning, within two hours after waking up, to account for the natural rise in cortisol levels during this time. We aim to collect these samples preferably between 6:30 AM and 8:30 AM.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Unger, MD, Principal Investigator — Sinai Health; Deborah O'Connor, PhD, RD, Study Director — Chair, Department of Nutritional Sciences, University of Toronto
Locations (3):
- Canada (3):
  - Labour and Delivery at Mount Sinai Hospital, Toronto, Ontario
  - Maternal Fetal Medicine and Placenta clinics, Toronto, Ontario
  - Placenta Clinic, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
All information collected during this study, including individual participant's personal health information, will be kept confidential and will not be shared with anyone outside the study unless required by law. Participants will not be named in any reports, publications, or presentations that may come from this study.

REFERENCES:
- [Background] Victora CG, Bahl R, Barros AJ, Franca GV, Horton S, Krasevec J, Murch S, Sankar MJ, Walker N, Rollins NC; Lancet Breastfeeding Series Group. Breastfeeding in the 21st century: epidemiology, mechanisms, and lifelong effect. Lancet. 2016 Jan 30;387(10017):475-90. doi: 10.1016/S0140-6736(15)01024-7. PMID 26869575
- [Background] Dennis CL, Brown HK, Chung-Lee L, Abbass-Dick J, Shorey S, Marini F, Brennenstuhl S. Prevalence and predictors of exclusive breastfeeding among immigrant and Canadian-born Chinese women. Matern Child Nutr. 2019 Apr;15(2):e12687. doi: 10.1111/mcn.12687. Epub 2018 Oct 4. PMID 30194811
- [Background] Vehling L, Chan D, McGavock J, Becker AB, Subbarao P, Moraes TJ, Mandhane PJ, Turvey SE, Lefebvre DL, Sears MR, Azad MB. Exclusive breastfeeding in hospital predicts longer breastfeeding duration in Canada: Implications for health equity. Birth. 2018 Dec;45(4):440-449. doi: 10.1111/birt.12345. Epub 2018 Mar 2. PMID 29498088
- [Background] Belfort MB, Drouin K, Riley JF, Gregory KE, Philipp BL, Parker MG, Sen S. Prevalence and Trends in Donor Milk Use in the Well-Baby Nursery: A Survey of Northeast United States Birth Hospitals. Breastfeed Med. 2018 Jan/Feb;13(1):34-41. doi: 10.1089/bfm.2017.0147. Epub 2017 Oct 24. PMID 29064280
- See also: Here is the link to the MaxiMOM (Maximizing Mothers Milk for Preterm Babies) studies, of which the CanDo trial is a part. — https://www.maximom-research.com/copy-of-research